CLINICAL TRIAL: NCT03738735
Title: Prospective, Double Blinded, Randomized Control Trial on Effect of Hyperosmlar Saline in Reducing Postoperative Pain Following Arthroscopic Rotator Cuff Repair
Brief Title: Randomized, Controlled Trial of Hyperosmotlar Saline for Rotator Cuff Repair Irrigation Solution
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018Davis
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Arthroscopic Shoulder Surgery; Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients will receive standard of care lactated ringer's solution for the arthroscopic irrigation during surgery.
- Intervention (Experimental): Patients will receive hyperosmolar saline for the arthroscopic irrigation during surgery.
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Hypertonic saline — For the intervention group, the surgical staff will add 120 mL of 23.4% saline to the 3L bags of lactated Ringer's solution, and this new solution will be used for arthroscopic irrigation purposes throughout the rotator cuff repair surgery.
  Arms: Intervention

SUMMARY:
The goal of this project is to perform a randomized, double-blinded study investigating postoperative pain after arthroscopic rotator cuff using hyperosmolar saline as opposed to lactated ringer's solution (normal osmolarity) as arthroscopy irrigation solutions. Hyperosmolar saline is an irrigation solution with a higher concentration of solutes that will be used intraoperatively to washout the surgical field. It will be used in place of lactated ringer's solution, which has an osmolarity comparable to that of normal saline. This study will help determine whether or not postoperative pain from rotator cuff repair can be mitigated by altering the osmolarity of the intraoperative irrigation solution. This knowledge is significant because the postoperative pain can be intense, so much so that patients may depend on narcotics for pain relief. Consequently, this study may provide benefit by helping to find new ways to minimize the need for narcotics. The main hypothesis of this is study is that hyperosmolar saline will reduce perceived pain and narcotic use in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years of age

Patients undergoing arthroscopic rotator cuff repair of full thickness, one or two tendon tears

Exclusion Criteria:

Patients younger than 18 years of age

Patients who are pregnant, mentally disabled, or imprisoned

Patients not receiving inter-scalene nerve block (catheters excluded)

Patients undergoing labral repair, capsular release, or distal clavicle excision

Patients with irreparable rotator cuff tears

Patients receiving any repair augmentation or graft

Patients with a known hypersensitivity to sodium lacta

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | daily for 14 days post-operatively
  pain rated on scale of 1-10
Morphine equivalent | weekly for first 2 weeks post-operatively
  opiod comsumption

SECONDARY OUTCOMES:
American Shoulder Elbow Surgeons standardized shoulder assessment form | 3 months and 6 months
  shoulder function
Passive range of motion | 6 weeks, 3 months, 6 months
  passive range of motion
Active range of motion | 3 months, 6 months
  Active range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Cox, MD, Principal Investigator — Thomas Jefferson University; Daniel Davis, MD, Study Director — Rothman Orthopaedics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capito NM, Cook JL, Yahuaca B, Capito MD, Sherman SL, Smith MJ. Safety and efficacy of hyperosmolar irrigation solution in shoulder arthroscopy. J Shoulder Elbow Surg. 2017 May;26(5):745-751. doi: 10.1016/j.jse.2017.02.021. Epub 2017 Mar 18. PMID 28318850
- [Background] Capito NM, Smith MJ, Stoker AM, Werner N, Cook JL. Hyperosmolar irrigation compared with a standard solution in a canine shoulder arthroscopy model. J Shoulder Elbow Surg. 2015 Aug;24(8):1243-8. doi: 10.1016/j.jse.2014.12.027. Epub 2015 Feb 25. PMID 25725966